CLINICAL TRIAL: NCT00463190
Title: Postmarketing Study of Probiotics Medication in Childhood Diarrhea
Brief Title: Effect of Probiotics (Bio-Three) in Children's Enterocolitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: X-BIO-440021
Record Dates: First submitted 2007-04-18; First posted 2007-04-20 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2007-04

CONDITIONS: Diarrhea; Enteritis; Enterocolitis
Keywords: Probiotics; Diarrhea; Enterocolitis
MeSH Terms: conditions — Diarrhea; Enteritis; Enterocolitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Biothree

SUMMARY:
Probiotic bacteria inhabit the gastrointestinal tracts of healthy individuals and may improve the health status of patients with digestive disease. The first aim of our study will seek to determine if probiotics medication (Bio-Three) inhibit gastrointestinal infection and reduce its inflammatory response in the intestine. The second aim will explore the bacterial count (microbiology) and subsequent immune response in probiotic inhibition of enterocolitis in children. We try to seek to gain an advanced understanding of probiotics versus pathogenic microorganism and host interactions, and mucosal immune responses to probiotics in the intestine.

DETAILED DESCRIPTION:
Viral infection is a leading cause of diarrhea in childhood . Rotavirus is the most common virus cause diarrhea among children worldwide. Probiotics are considered to be beneficial in the management and prevention of viral diarrhea. Saavedra et al. had reported that feeding an infant formula with Streptococcus thermophilus and Bifidobacterium bifidum can reduce the incidence of diarrhea and rotavirus shedding in infants. Another study suggests that children receiving a bifidobacteria-supplemented milk-based formula may be protective against symptomatic rotavirus infection.

Several pathogens, such as Salmonella spp., enteropathogenic Escherichia coli and enterohemorrhagic E. coli spp., Campylobacter spp., Shigella spp., can cause invasive diarrhea. These pathogens have the capacity to invade the mucosa of the distal small intestine and colon, stimulate local and systemic inflammatory responses, and sometimes causing hemorrhage and ulceration of the mucosa. Some strains of invasive bacteria not only induce intestinal cellular damage but also enter the systemic circulation to affect distal organs. Probiotics have been shown to be effective in the treatment of these conditions. There are many mechanisms by which probiotics enhance intestinal health, including stimulation of immunity, competition for limited nutrients, inhibition of epithelial and mucosal adherence, inhibition of epithelial invasion and production of antimicrobial substances .

Clostridium butyricum is effective for both the treatment and the prophylaxis of antibiotic-associated diarrhea in children, as it normalizes the intestinal flora disturbed by antibiotics. Probiotics ( Bacillus mesentericus) affect intestinal bacterial flora by increasing anaerobic bacteria and decreasing the population of potentially pathogenic microorganisms. A decrease in luminal endotoxin may result in less endotoxin translocation or bacterial translocation. The effect of Bio-Three (Enterococcus T-110, C. butyricum TO-A, B. mesentericus TO-A) was ever proved on (a) normalization of enterobacterial flora, (b) improvement of growing abilities of live bacteria in the drug, (c) inhibition of pathogenic bacteria , (d) promotion of the growth of beneficial bacteria . Despite the gastrointestinal effect, Bio-three therapy was also effective in both clinical and bacteriological responses in genital tract infection by published literature.

ELIGIBILITY:
Inclusion Criteria:

* Clinical symptom of diarrhea less than 3 days

Exclusion Criteria:

* Severe abdominal distension with risk of bowel perforation
* Risk for sepsis
* Past history with surgical operation of gastrointestinal tracts

Ages: 3 Months to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2006-02; Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Clinical symptom 2 days after medication
Microbiology study 3 days and one week after medication

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chang Chen, MD, Principal Investigator — Pediatrics, Chang Gung Memorial Hospital & Chang Gung University College of Medicine & Chang Gung Children's Hospital
Locations (1):
- Pediatrics, Chang Gung Memorial Hospital & Chang Gung University College of Medicine & Chang Gung Children's Hospital, Taoyuan District, Taiwan

REFERENCES:
- [Background] Chen CC, Walker WA. Probiotics and prebiotics: role in clinical disease states. Adv Pediatr. 2005;52:77-113. doi: 10.1016/j.yapd.2005.03.001. PMID 16124337
- [Derived] Chen CC, Kong MS, Lai MW, Chao HC, Chang KW, Chen SY, Huang YC, Chiu CH, Li WC, Lin PY, Chen CJ, Li TY. Probiotics have clinical, microbiologic, and immunologic efficacy in acute infectious diarrhea. Pediatr Infect Dis J. 2010 Feb;29(2):135-8. doi: 10.1097/inf.0b013e3181b530bf. PMID 20135748
- See also: Click here — http://www.cgmh.org.tw/